CLINICAL TRIAL: NCT03422913
Title: Controlled Low Central Venous Pressure Combined With Hilar Block in Laparoscopic Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2017-073-01
Record Dates: First submitted 2018-01-10; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopic Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both patients and surgeons are blinded, and anesthesiologist opened the envelope during the operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLCVP Group (Experimental): Controlled low central venous pressure(CLCVP) will be performed combined with intraoperative combined hilar intermittent (Pringle method)
  Interventions: Procedure: controlled low central venous pressure
- Control Group (No Intervention): Only intraoperative combined hilar intermittent (Pringle method) will be performed

INTERVENTIONS:
Procedure: controlled low central venous pressure — Anesthesiologists will control the amount of fluid input and the use of composite intravenous anesthesia to make CVP at 0~5cm H2O, if CVP is still >5cm H2O, intravenous infusion of nitroglycerin will be used to reduce CVP. Maintaining arterial systolic blood pressure (SBP) > 90 mmHg, urine output more than 1ml/kg/h, and CVP was continuously monitored. Arterial pressure, pulse oxygen saturation ( SPO2), PaCO2 and electrocardiogram (II and V5 leads) were continuously monitored by radial artery cannulation. CVP will Returned to normal level (6 ~ 12 cmH2O) after resection to observe the wound if active bleeding still exist. Intraoperative hepatic blood flow blocking intermittent Pringle block method also required during surgery, 10-15 minutes for once, and more than 5 minutes interval can be repeated.
  Arms: CLCVP Group

SUMMARY:
Hepatectomy is the preferred method for the treatment of liver tumors. Since the liver is a double blood supply organ, massive hemorrhage during hepatectomy may lead to hemodynamic instability, prolonged portal vein occlusion and increased ischemia-reperfusion injury. In addition, bleeding during hepatectomy, intraoperative and postoperative blood transfusion are the main causes of postoperative morbidity and mortality. Therefore, bleeding control during liver resection is a critical technique. Based on the fact that liver is more tolerant to warm ischemia and hypoxia, a variety of techniques have been widely used for hepatic blood flow occlusion.

With the prevalence of laparoscopy, more patients received laparoscopic resection of liver cancer. Bleeding has become a major constraint, so how to reduce the bleeding and preserve liver function has always been surgeons' concern.As conventional hepatic portal blood flow blocking technology is more mature, the risk of bleeding during laparoscopic liver resection mainly comes from hepatic veins in the process of hepatic parenchymal isolation. Although Ultrasound scalpel and Ligasure have been widely accepted in the treatment of laparoscopic hepatectomy, due to the thin hepatic vein and the high intraluminal pressure, it is also difficult to control the bleeding during surgery. How to prevent hepatic venous hemorrhage has become the key to reduce the bleeding . As sinusoidal pressure is affected by intrahepatic pressure, which is directly related to central venous pressure (CVP), reducing CVP can reduce the pressure in the hepatic veins and sinusoids hence reducing bleeding when the hepatic parenchyma is severed. That is the rationale of controlled low central venous pressure CLCVP) to reduce the risk of hepatectomy, which have been used maturely in open hepatectomy. Due to the low risk of hepatic and renal insufficiency and gas embolism in liver surgery, there is a potential risk of laparoscopic pneumoperitoneum and the risk of laparoscopic pneumoperitoneum is further increased. Therefore, how to implement CLCVP in laparoscopic surgery to reduce the risk of bleeding, also avoiding complications such as bleeding gas embolism, is a clinical problem to be solved, is rarely reported. A prospective randomized controlled trial (RCT) will be performed for laparoscopic hepatectomy in patients combine intraoperative combined hilar intermittent (Pringle method) with or without CLCVP to reduce the bleeding. This study was to investigate the safety and efficacy of CLCVP in combination with intermittent Pringle.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis or pathological diagnosis of hepatocellular carcinoma;
2. resectable non-left lobes, left and right liver lesions, and the resection range is expected to be greater than or equal to 1 liver segment, no non-cancerous thrombus; Indocyanine Green Retention Rate (ICGR) 15 minutes retention rate <10%
3. did not receive systemic chemotherapy or other targeted drug therapy for diagnosing hepatocellular carcinoma(HCC) before participating in the study;
4. generally good, Karnofsky Performance Scores (KPS) ≥ 80 points;
5. Age: 18-70 years old
6. Child-Pugh A level
7. Baseline laboratory tests meet the following criteria:

white blood cells ≥ 3.0 × 109 / L platelets ≥ 75 × 109 / L hemoglobin ≥ 100g / L serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) serum creatinine ≤ 1.5 x ULN International normalized ratio （INR）<1.4, or prothrombin time <ULN + 4 seconds albumin ≥ 30g / L Total bilirubin ≤34mmol / L

Exclusion Criteria:

1. patients do not agree to participate in clinical studies;
2. Any of the following had been reported in the 12 months prior to participating in the study: myocardial infarction, severe / unstable angina, coronary artery bypass surgery, congestive heart failure, cerebrovascular accident (including transient ischemic attack), Pulmonary Embolism; Ongoing: corrected QT interval prolongation (≥450 ms for males and> 470 ms for females) according to NCI-CTCAE criteria ≥2 arrhythmias;
3. There are other serious acute and chronic physical or mental illnesses or laboratory abnormalities that may increase the risk associated with participating in study treatment or may interfere with the interpretation of the findings or in patients deemed inappropriate by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | During surgery procedure
  Blood loss in the two treatment groups were compared.

SECONDARY OUTCOMES:
Safety | During surgery procedure
  Incidence of gas embolism caused transient hypoxemia
Liver function recovery | within 5 days after surgery
  blood test to show liver function recovery after surgery, that is elevation of transaminase

CONTACTS AND LOCATIONS:
Overall Officials: Zhongguo Zhou, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pan YX, Wang JC, Lu XY, Chen JB, He W, Chen JC, Wang XH, Fu YZ, Xu L, Zhang YJ, Chen MS, Lai RC, Zhou ZG. Intention to control low central venous pressure reduced blood loss during laparoscopic hepatectomy: A double-blind randomized clinical trial. Surgery. 2020 Jun;167(6):933-941. doi: 10.1016/j.surg.2020.02.004. Epub 2020 Mar 23. PMID 32216964